CLINICAL TRIAL: NCT01059110
Title: Comparison of Occlusive Dressings, Salicylate Ointment, Cryotherapy, Topical 5-fluoro-uracil and Imiquimod in Immunocompetent Patients Presenting Plantar Warts in Office-based Settings: a Randomized Clinical Trial
Brief Title: Comparison of Five Treatments in Patients With Plantar Warts
Acronym: VRAIE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty to enrollment patients
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Society of Dermatology and venerology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070701
Record Dates: First submitted 2009-11-30; First posted 2010-01-29 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Plantar Warts
Keywords: Occlusive dressings; Salicylate ointment; Cryotherapy; Topical 5-fluoro-uracil; Imiquimod; Randomized clinical trial; Plantar warts
MeSH Terms: interventions — Imiquimod; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Salicylate ointment (Experimental): Salicylate ointment under occlusion (pomade M.O Cochon®)
  Interventions: Drug: Salicylate ointment
- Imiquimod (Experimental): Imiquimod : Aldara®
  Interventions: Drug: Imiquimod
- 5-fluoro-uracil (Experimental): 5-fluoro-uracil cream : Efudix®
  Interventions: Drug: 5-Fluoro-Uracil
- Cryotherapy (Experimental): liquid nitrogen : Cryotherapy
  Interventions: Drug: Cryotherapy

INTERVENTIONS:
Drug: Salicylate ointment — cream, one application every night, for 90 days
  Other Names: pommade M.O Cochon®
  Arms: Salicylate ointment
Drug: Imiquimod — cream, one dose of 250 mg, one application 3 times a week during 12 hours, for 90 days
  Other Names: Aldara® 5%
  Arms: Imiquimod
Drug: 5-Fluoro-Uracil — cream, one application every night, during 12 hours, for 90 days
  Other Names: Efudix® 5%
  Arms: 5-fluoro-uracil
Drug: Cryotherapy — 2 cycles of 5 seconds after obtention of halo of white
  Other Names: Liquid nitrogen
  Arms: Cryotherapy

SUMMARY:
The principal objective of the study is to compare 5 usual strategies in the management of plantar warts which did not cure after 5 weeks of a salicylate ointment given just prior the trial. The trial will include immunocompetent patients coming from the community and should help the office-based dermatologists and hospital in the decision-making therapeutic process.

DETAILED DESCRIPTION:
Four and a half million individuals in France have warts (SOFRES poll 2002). Notably, plantar warts are considered to be the most common reason for consulting a private practitioner, despite the absence of robust epidemiological data. Although benign, plantar warts are associated with a certain degree of morbidity: pain, difficulty walking, and intra- and interindividual contagion. Despite the frequency of plantar warts and patients high expectations for their treatments, which are numerous for immunocompetent patients, those remedies have only been evaluated in undeniably inadequate ways. Patient demand for therapy is strong, with those affected going from one physician to another, in the search for the "good treatment". For all the reasons evoked in the context of skin diseases, healing warts can indeed represent a public health objective.

One of the difficulties of evaluating treatments is the frequency of spontaneous complete remissions (natural history) and/or under placebo, assessed at 30% [range: 0-73%] in a short-term trial (10 weeks). In addition, professionals experiences support frequent relapses that have been very poorly evaluated in therapeutic trials.

Keratolytic treatment, usually salicylated petroleum jelly, is the standard therapy according to the Cochrane Review. In practice, this therapy usually combines manual shaving, done by the patient him/herself or the physician. Supplementing this basic therapy with a physical (standard cryotherapy), chemical (5-fluorouracil; Efudix®) or immunological adjunct (imiquimod; Aldara®), to achieve the desired effect of increasing the frequency and/or rapidity of complete cure, has never been examined in a large randomized-controlled trial.

A population comprised of patients with warts still "resistant" after 5 weeks of keratolytic therapy with 50% salicylic acid (PommadeM.O Cochon®) followed by a 1-week washout was deliberately retained because it is this precise setting that poses therapeutic difficulties in routine practice. The 1-week washout will allow the skin to heal a little and facilitate the diagnosis of failures; and, moreover, the strategy of pretreatment with scraping would not be unduly weakened.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 years or more.
* Clinical evaluation
* Number of warts lower than 10 on the 2 feet and total diameter of warts lower than 10 cm, whether previously treated or not
* In treated patients, all potentially active treatment on warts since at least one month should be stopped.
* Effective contraception for women of childbearing age
* Immunocompetent patients
* Patient with one or more warts on soles and board feet.

  * MYRMECIE : rounded warts, deep, covered with a stratum corneum more or less thick; after stripping, appear black points, very specific; often painful to pressure. They are lonely, single or not. They could regroup galley thick. The stripping can them to individualize.
  * Mosaic : plate small warts, superficial, often sitting on the heel or Forefoot. Little painful, they are often ignored by the patients when they appear
* Patient affiliated to the French social security.

Exclusion Criteria:

* Patient suspected to be immunocompromised
* Patient aged under 18 years
* Patient refusing to sign the consent
* Pregnant or lactating women
* Plantar calluses
* Known hypersensitivity to imiquimod (Aldara®) or any excipients of the cream (isostearic acid, benzyl alcohol, cetyl alcohol, stearyl alcohol, paraffin, polysorbate 60, sorbitan stearate, glycerol, methyl hydroxybenzoate, propyl hydroxybenzoate, xanthan gum, purified water)
* Known hypersensitivity to 5 fluoro-uracil (Efudix®) or any excipients of gel (stearyl alcohol, Vaseline, polysorbate 60, propyleneglycol, purified water - conservatives: METHYL PARAHYDROXYBENZOATE, PROPYL PARAHYDROXYBENZOATE)
* Contra-indication to Pomade M.O Cochon® (Known allergy to any components)
* Known hypersensitivity to Blenderm®
* Extra plantar concomitant warts (to exclude risk of endogenous recontamination by an extra plantar site)
* Plantar hyperhidrosis making impossible adhesion of plaster.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2010-02; Primary Completion 2015-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Complete clinical remission of the warts assessed by the dermatologist | at 90 days

SECONDARY OUTCOMES:
Time remission | at 30, 60 and 90 days
Number of warts in remission vs baseline | at 30, 60 and 90 days
Time to first relapse | at 30, 60, 90, 120, 180, 360 and 720 days
Percentage of relapse (phone call assessment) | at 360 days and 720 days
Safety | at 90 days
Evaluation of distress (visual analogic scale) | at 90 days
Compliance. | at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHOSIDOW, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Medical center, Athis-Mons, France

REFERENCES:
- [Derived] Chanal J, Aubin F, Penso-Assathiany D, Buffiere I, Makhlouf W, Perriere C, Bocquet H, Aubin A, Farcet Y, Ludmann C, Duboz A, Marco-Bonnet J, Maury C, Tremeau-Martinage C, Hubert-Asso AM, Coustou D, Heudes AM, Kemula M, Beylot-Barry M, Tetart F, Eche-Dejoie A, Duvochel AM, Baspeyras M, Amici JM, Toussaint H, Neculaita L, Mboup B, Pizzi N, Jouis V, Vacher Y, Pretet JL, Vicaut E, Chosidow O. A multicentre pragmatic randomized controlled trial comparing 50% salicylic acid, liquid nitrogen, 5% 5-fluorouracil cream, and 5% imiquimod cream in previously treated plantar warts. The VRAIE (VeRrues plAntaIres en villE) study. Ann Dermatol Venereol. 2025 Sep;152(3):103406. doi: 10.1016/j.annder.2025.103406. Epub 2025 Jul 30. PMID 40743833